CLINICAL TRIAL: NCT06816615
Title: Diagnosis and Percutaneous Treatment of Biliary Tract Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPY2021
Record Dates: First submitted 2025-01-09; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Gallstone; Biliary Stricture; Biliary Diseases
MeSH Terms: conditions — Gallstones; Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with bile duct disease not eligible for endoscopic treatment (Experimental): Before the procedure all patients will be submitted to US and/or CT and/or MRI and will be evaluated for hemoglobin, hematocrit and liver function tests. Patients with biliary tract disorders that are not eligible for endoscopic treatment and/or previous failed endoscopic treatment will be evaluated for inclusion in this study. Therefore, a case-by-case discussion will be conducted with the reference hepatologists/surgeons to assess treatment assignment. Once enrolled in the study, patients will undergo cholangioscopic-assisted treatment at the UOC addomino-pelvic diagnostic and interventional radiology unit of the Bologna University Hospital. After the procedure, patients will be required to perform a clinical laboratory monitoring in subsequent follow-up controls that will be performed 3-6-12-24-36 months after treatment. Additional imaging examinations (US, CT or MRI) will only be scheduled if symptoms recur.
  Interventions: Procedure: Percutaneous cholangioscopic-assisted treatment

INTERVENTIONS:
Procedure: Percutaneous cholangioscopic-assisted treatment — The intervention administered is a percutaneous colangioscopic assisted technique that uses endoscopic Spyglass system. The endoscopic Spyglass system is designed to provide direct viewing and to guide both optical devices and accessories for lithotripsy in case of litiasic pathology and is equipped with a suitable bioptic clamp in case of biopsy collection. The use of the digital Spyglass catheter involves the preliminary percutaneous puncture of the bile ducts with a right, left or combined approach, and the subsequent execution of a cholangiographic study. Additional treatment sessions may be performed every 15-20 days in case of residual lithiasis. At the end of each session, an internal-external transeptic percutaneous drainage (ptbd) of adequate caliber (8-14 fr) is left in place to monitor any complications and maintain a route of access for sequential treatments.

SUMMARY:
This study aims to implement and optimize the treatment of bile duct diseases in participants not eligible for endoscopic treatment using the Spyglass system, a system suitable for diagnostic and therapeutic endoscopic procedures in the pancreatic-biliary system, including the hepatic ducts.

The main question it aims to answer is:

- Can the percutaneous cholangioscopic assisted technique resolve the biliary litiasis and/or perform endobiliary biopsies in less time than the traditional technique?

Participants will undergo a colangioscopic-assisted treatment using the SpyGlass mini-endoscopic system at the Addomino-pelvic diagnostic and interventional radiology UOC of the Bologna University Hospital.

DETAILED DESCRIPTION:
This is a pilot, spontaneous, non-pharmacological, prospective and single-center interventional study aimed at participants with bile duct diseases not eligible for endoscopic treatment, who, once enrolled, will undergo percutaneous colangioscopic-assisted treatment at the Addominal-pelvic diagnostic and interventional radiology UOC of the University Hospital of Bologna. After a 24-month enrollment phase, a 36-month follow-up phase will be undertaken to assess the functional and therapeutic outcomes of this approach.

The enrollment and the collection of informed consent will be carried out by the Radiologists involved in the study who will also take care of the collection of clinical data and the review of all pseudoanymous radiological images pre/post treatment in order to evaluate the outcome of percutaneous treatment, the number of treatments, the duration of drainage stay, the relapse-free interval and the length of hospitalization. Participants in the study will undergo treatments commonly used in daily clinical practice, including biliary clearance and/or endobiliary biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of indeterminate gallstones or stenosis of the bile ducts not eligible for endoscopic treatment and/or previous failed endoscopic treatment
* Good liver function (hemoglobin, hematocrit, GOT, GPT, GGT within normal ranges)
* Age over 18
* Obtaining informed consent

Exclusion Criteria:

* presence of severe untreatable coagulopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of treatments | From enrollment to the end of treatment at 7 years
  Number of treatments
Duration of drainage | From enrollment to the end of treatment at 7 years
  Duration of drainage
Relapse free interval | From enrollment to the end of treatment at 7 years
  Relapse free interval
Duration of hospitalization | From enrollment to the end of treatment at 7 years
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Alberta Cappelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy